CLINICAL TRIAL: NCT03912792
Title: A Cross-Sectional Natural History Study to Evaluate Sweat Volume and Other Phenotypic and Genetic Characteristics in Patients Affected by X-Linked Hypohidrotic XLHED Ectodermal Dysplasia (XLHED)
Brief Title: A Cross-Sectional Natural History Study to Evaluate Sweat Volume and Other Phenotypic and Genetic Characteristics in Patients Affected by XLHED
Status: Withdrawn | Type: Observational
Why Stopped: Company decision
Sponsor: Dermelix Biotherapeutics, LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: DMX101-0001
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: XLHED
Keywords: Natural History Study; X-Linked Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

GROUPS / COHORTS (2):
- XLHED Patients
- Healthy Controls

SUMMARY:
The proposed natural history study will enroll male patients with a diagnosis of XLHED, female carriers of XLHED and healthy volunteers. The study protocol will include collection of XLHED questionnaires and clinical outcomes using minimally invasive technologies. Data will be collected both retrospectively and prospectively.

Clinical outcome assessments will be performed at the NFED Family Conference on July 11-12, 2019. Study participants will be able to complete XLHED questionnaires electronically ahead of the conference.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Males with XLHED, female carriers of XLHED and healthy volunteers

Exclusion Criteria:

* Treatment with an investigational study drug for XLHED
* Any major medical problems that would prevent her/him from participating in this study
* Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists (Examples: Urecholine, Salagen, Pilocar, and Provocholine)
* Pacemaker

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Males with XLHED and female carriers of XLHED
  Male and female healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The volume of sweat from a pilocarpine-induced sweat test | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Chicago Marriott Lincolnshire Resort, Lincolnshire, Illinois, United States